CLINICAL TRIAL: NCT00913107
Title: Lamotrigine in Trigeminal Neuralgia: Efficacy and Safety in Comparison With Carbamazepine
Brief Title: Efficacy and Safety Study of Lamotrigine to Treat Trigeminal Neuralgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Dr. Sameer Shaikh, Dept. of OMOP, Faculty of Dentistry, University Malaya.
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PS287-2007B
Record Dates: First submitted 2009-05-27; First posted 2009-06-03 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; Lamotrigine; Carbamazepine; Lamictal®; Tegretol®
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lamotrigine; Carbamazepine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamictal® (Experimental): Lamictal® was used as the "active" medication in this study.
  Interventions: Drug: Lamictal®; Drug: Tegretol®
- Tegretol® (Active Comparator): Tegretol® was employed as the "control" for comparative purposes in order to check and evaluate the efficacy (pain-relief) and occurrence of side- effects of Lamictal®.
  Interventions: Drug: Lamictal®; Drug: Tegretol®

INTERVENTIONS:
Drug: Lamictal® — The regime of prescription for Lamictal® during the clinical trials was as follows:
  1. 50 mg twice daily for 10days, followed by,
  2. 100 mg twice daily for the next 10days, followed by,
  3. 100 mg thrice daily for the next10 days, followed by,
  4. 100 mg four times daily for the final 10 days.
  Other Names: Lamotrigine (generic name for Lamictal®); Carbamazepine (generic name for Tegretol®)
Drug: Tegretol® — The regime of prescription for Tegretol® during the clinical trials was as follows:
  1. 150 mg twice daily for 10days, followed by,
  2. 200 mg thrice daily for the next 10days, followed by,
  3. 300 mg thrice daily for the next 10 days, followed by,
  4. 300 mg four times daily for the final 10 days.
  Other Names: Lamotrigine (generic name for Lamictal®); Carbamazepine (generic name for Tegretol®)

SUMMARY:
The purpose of this study was to determine the efficacy and safety of lamotrigine in patients with trigeminal neuralgia (TGN).

DETAILED DESCRIPTION:
Trigeminal Neuralgia (TGN) is a rare form of chronic facial pain shrouded in mystery, although not life threatening, can be excruciating painful and extraordinarily debilitating. Its uniqueness and peculiarity can be ascertained by the fact that TGN may present to and be managed by dentists, neurologists, neurosurgeons, oral surgeons and ear, nose and throat surgeons.

The management of TGN is initially medical, with the "gold standard" drug of carbamazepine (CBZ). Whilst CBZ continues to be the treatment of choice, a substantial proportion of patients tolerate this drug poorly, predominantly because of side-effects that include drowsiness, accommodation disorders, hepatitis, elevation in liver enzymes, renal dysfunction, congestive heart failure, delayed multi-organ failure, leucopenia, thrombocytopenia etc. etc. If pain-relief is incomplete with CBZ or it produces adverse side-effects, options include using an alternative second-line medical agent. The drugs suggested to be considered as second-line agents for the treatment of TGN, include: lamotrigine, baclofen, phenytoin, oxcarbazepine, gabapentin, clonazepam, valproate, mexiletine, and topiramate.

Lamotrigine (LTG), a novel anticonvulsant, which has not been adequately assessed for its antineuralgic properties. It has a bimodal mechanism of action:

* inhibits the release of glutamate and aspartate by blocking voltage-sensitive sodium channels
* antagonistic at neuroexcitatory N-methyl-d-aspartate receptors.

It can also acts at and inhibits calcium channels to enhance the gamma- Aminobutyric acid (GABA) synthesis. GABA is an inhibitory amino acid neurotransmitter that decreases neural membrane action potentials and therefore decreases nerve excitability. Glutamate has been implicated in the mechanisms contributing towards phenomenon of chronic pain, such as sensitisation and wind up. LTG through its inhibition of pathological release of glutamate, has the potential towards management of chronic pain, particularly of neuropathic origin.

Lamotrigine, therefore has the potential to be a promising new treatment for TGN.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Trigeminal Neuralgia
* Male; or non-pregnant/non-lactating female
* Must be willing to cooperate with and understands study instructions
* Signed informed consent prior to entering study

Exclusion Criteria:

* psychiatric illness
* severe liver or cardiovascular disease
* renal impairment, low white cell count
* malignancy
* pregnancy or lactation
* alcohol or recreational drug abuse
* and positive tests for human immunodeficiency virus or hepatitis B or C.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pain-relief | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sameer Shaikh, MDSc., Principal Investigator — Faculty of Dentistry, University Malaya
Locations (2):
- Malaysia (2):
  - Dept. of OMOP, Faculty of Dentistry, University Malaya., Kuala Lumpur
  - Dept. of Oral Medicine and Oral Pathology, Faculty of Dentistry, University Malaya., Kuala Lumpur

REFERENCES:
- [Derived] Shaikh S, Yaacob HB, Abd Rahman RB. Lamotrigine for trigeminal neuralgia: efficacy and safety in comparison with carbamazepine. J Chin Med Assoc. 2011 Jun;74(6):243-9. doi: 10.1016/j.jcma.2011.04.002. Epub 2011 May 10. PMID 21621166